CLINICAL TRIAL: NCT01643421
Title: Effects of a Program of Deep Inspiration Combined to Expiratory Positive Airway in Quality of Life and Heart Rate Variability
Brief Title: Effect of a Program of Deep Inspiration Combined to Expiratory Positive Airway Pressure in Asthmatic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Pedro Dal Lago, Professor, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: II+EPAP
Record Dates: First submitted 2012-07-10; First posted 2012-07-18 (Estimated); Last update posted 2014-08-11 (Estimated); Status verified 2014-08

CONDITIONS: Improvement of Functional Capacity.; Improvement of Quality of Life.; Improvement of Cardiovascular Autonomic Control.

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Deep inspiration and expiratory positive airway pressure (Experimental): The protocol of deep inspiration combined to expiratory positive airway pressure will be applied in asthmatic subjects.
  Interventions: Other: Deep inspiration and positive expiratory airway pressure
- Control (No Intervention)

INTERVENTIONS:
Other: Deep inspiration and positive expiratory airway pressure — It was used a device the combines deep inspiration and positive expiratory airway pressure in asthmatic subjects, for 5 weeks, twice a day.
  Arms: Deep inspiration and expiratory positive airway pressure

SUMMARY:
The purpose of this study is to determine the effects of a deep inspiration combined to expiratory positive airway pressure protocol on respiratory function, quality of life, exercise tolerance and heart rate variability in adults with severe asthma.

DETAILED DESCRIPTION:
Asthma is associated with high morbidity and significant mortality. This disease has functional impact on activities of daily living (ADLs) and according to some studies in the United States and Europe, the percentage of asthmatics who have significant restrictions in their ADLs is quite significant. Asthma is characterized as a major public health problem, not only in Brazil but worldwide. Currently there are few studies reporting the effects of a domiciliary program of deep inspiration associated with positive expiratory pressure in the airways of asthmatics. This study aims to analyze the benefits of this program on lung function, quality of life and response to exercise.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 80
* Severe asthma

Exclusion Criteria:

* Disagreement with consent form
* Other respiratory disease
* Acute severe asthma
* Pregnancy or breastfeeding
* Current smoking
* Lack of capable of conducting the study visits

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-01; Primary Completion 2012-05 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
The effect of deep inspiration and positive expiratory airway pressure in quality of life in adults with severe asthma | Change in quality of life at 5 week
  The quality of life will be measure by a specific questionnaire for this population 5 weeks apart.

SECONDARY OUTCOMES:
The effect of deep inspiration and positive expiratory airway pressure in respiratory function in adults with severe asthma. | Change in respiratory function at 5 week
  The respiratory function will be measure by spirometry 5 weeks apart.
The effect of deep inspiration and positive expiratory airway pressure in heart rate variability in adults with severe asthma. | Change in heart rate variability at 5 week
  The heart rate variability will be measure by the acquisition of electrocardiogram signal 5 weeks apart.
The effect of deep inspiration and positive expiratory airway pressure in exercise tolerance in adults with severe asthma. | Change in exercise tolerance at 5 week
  The exercise tolerance will be measure by 6 minute walk test 5 weeks apart.

CONTACTS AND LOCATIONS:
Locations (1):
- Pedro Dal Lago, Porto Alegre, Rio Grande do Sul, Brazil